CLINICAL TRIAL: NCT06765083
Title: Can We 'hear' Femoral Neck Fractures? Ultrasound Guided Diagnosis of Femoral Neck Fractures.
Acronym: CHEFF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Frisius Medisch Centrum (Other)
Responsible Party: Principal Investigator, Svenja Haak, MD, Frisius Medisch Centrum
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 202400397
Record Dates: First submitted 2024-12-03; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Hip Fractures (i.e. Femoral Neck or Intertrochanteric Hip Fractures)
Keywords: femoral neck; pertrochanteric; hip; fracture; POCUS; ultrasound; diagnostic; Emergency Department; proximal femur
MeSH Terms: conditions — Hip Fractures; Fractures, Bone; Disease; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- All participants (Experimental): All patients enrolled in the study will undergo POCUS of the hip by the (resident) emergency physician, prior to radiograph imaging.
  Interventions: Diagnostic Test: POCUS of the hip

INTERVENTIONS:
Diagnostic Test: POCUS of the hip — POCUS of the hip (proximal femur) by the (resident) emergency physician, prior to radiograph imaging.

SUMMARY:
Hip (femoral neck and pertrochanteric) fractures account for a significant part of Emergency Department (ED) visits after trauma. Studies suggest that point-of-care ultrasound (POCUS) is a reliable diagnostic tool for fracture assessment. POCUS has several advantages over conventional radiography, such as being portable, cheaper and radiation free. In addition, immediate conversion to ultrasound guided regional anaesthesia upon diagnosis of fracture can improve patient's time to proper analgesia. Moreover, POCUS can potentially be used pre-hospital to rule out hip fractures reducing ED crowding, as well as being a solution for areas where radiography is not readily available (e.g. rural or developing areas).

The primary objective of this study, is to evaluate the diagnostic capabilities of POCUS regarding patients with suspected hip fracture after trauma compared to radiography, the current standard of care diagnostic tool.

DETAILED DESCRIPTION:
Rationale: Hip (femoral neck and pertrochanteric) fractures account for a significant part of Emergency Department (ED) visits after trauma. Studies suggest that point-of-care ultrasound (POCUS) is a reliable diagnostic tool for fracture assessment. POCUS has several advantages over conventional radiography, such as being portable, cheaper and radiation free. In addition, immediate conversion to ultrasound guided regional anaesthesia upon diagnosis of fracture can improve patient's time to proper analgesia. Moreover, POCUS can potentially be used pre-hospital to rule out hip fractures reducing ED crowding, as well as being a solution for areas where radiography is not readily available (e.g. rural or developing areas).

Objective: Our primary objective is to evaluate the diagnostic capabilities of POCUS regarding patients with suspected hip fracture after trauma compared to radiography, the current standard of care diagnostic tool.

Study design: Prospective cohort study. Study population: All patients aged 18 and older presenting to the ED with a painful hip after trauma suspected of hip fracture are eligible to be enrolled in this study.

Intervention: Patients enrolled in the study will undergo POCUS of the hip (femoral neck) by the (resident) emergency physician, prior to radiograph imaging.

Main study parameters/endpoints: Sensitivity, specificity, positive predicting value (PPV) and negative predicting value (NPV) of POCUS in detecting hip fractures by assessing for posttraumatic changes (cortical disruptions, joint effusion and peritrochanteric edema).

Informed consent will be requested and documented.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* presenting to the ED with a painful hip after trauma, suspected of hip fracture as defined by the attending clinician

Exclusion Criteria:

* History of hip fracture or surgical procedure on the bones of the ipsilateral hip (ultrasound images may be unreliable)
* Presence of foreign body material in the ipsilateral hip
* Skin defects at the POCUS site e.g. lacerations, infected skin
* Extensive injuries, extreme pain or neurovascular damage where urgent intervention is required
* Inability to give informed consent (cognitive impairments, no proficient understanding of the Dutch or English language)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of POCUS | From enrollment to the end of POCUS, approximately 10 to 30 minutes
  Diagnostic accuracy (sensitivity, specificity, negative predicting value (NPV) and positive predicting value (PPV)) of POCUS in detecting hip fractures by assessing for posttraumatic changes (cortical disruptions, joint effusion and peritrochanteric edema).

SECONDARY OUTCOMES:
Difference in diagnostic accuracy of POCUS in diagnosing a femoral neck or pertrochanteric fracture | From enrollment to the end of POCUS, approximately 10 to 30 minutes
  Difference in diagnostic accuracy (sensitivity, specificity, negative predicting value (NPV) and positive predicting value (PPV)) of POCUS in diagnosing a femoral neck or pertrochanteric fracture
Difference in diagnostic accuracy of POCUS in detecting hip fractures stratified by operator experience (in years) using POCUS | From enrollment to the end of POCUS, approximately 10 to 30 minutes
  Difference in diagnostic accuracy (sensitivity, specificity, negative predicting value (NPV) and positive predicting value (PPV)) of POCUS in detecting hip fractures stratified by operator experience (in years) using POCUS
Difference in effusion measured in mm between the ipsilateral and contralateral hip | From enrollment to the end of POCUS, approximately 10 to 30 minutes
  Difference in effusion measured in mm between the ipsilateral and contralateral hip
Added value of POCUS in detecting hip fractures compared to the likelihood determined through clinical assessment by the treating physician | From enrollment to the end of POCUS, approximately 10 to 30 minutes
  Evaluate the added value of POCUS in detecting hip fractures compared to the likelihood determined through clinical assessment by the treating physician (questionnaire: hip fracture clinical suspected yes or no)

CONTACTS AND LOCATIONS:
Locations (1):
- Medisch Centrum Leeuwarden, Leeuwarden, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bossuyt PM, Reitsma JB, Bruns DE, Gatsonis CA, Glasziou PP, Irwig L, Lijmer JG, Moher D, Rennie D, de Vet HC, Kressel HY, Rifai N, Golub RM, Altman DG, Hooft L, Korevaar DA, Cohen JF; STARD Group. STARD 2015: an updated list of essential items for reporting diagnostic accuracy studies. BMJ. 2015 Oct 28;351:h5527. doi: 10.1136/bmj.h5527. PMID 26511519
- [Background] Koski JM, Anttila PJ, Isomaki HA. Ultrasonography of the adult hip joint. Scand J Rheumatol. 1989;18(2):113-7. doi: 10.3109/03009748909099926. PMID 2660254
- [Background] Cohen A, Li T, Greco J, Stankard B, Mingione P, Huang V, Gold A, Zarider N, Nutovits A, Nelson M. Hip effusions or iliopsoas hematomas on ultrasound in identifying hip fractures in the emergency department. Am J Emerg Med. 2023 Feb;64:129-136. doi: 10.1016/j.ajem.2022.11.034. Epub 2022 Dec 1. PMID 36521235
- [Background] Hajian-Tilaki K. Sample size estimation in diagnostic test studies of biomedical informatics. J Biomed Inform. 2014 Apr;48:193-204. doi: 10.1016/j.jbi.2014.02.013. Epub 2014 Feb 26. PMID 24582925
- [Background] Berg LM, Ehrenberg A, Florin J, Ostergren J, Discacciati A, Goransson KE. Associations Between Crowding and Ten-Day Mortality Among Patients Allocated Lower Triage Acuity Levels Without Need of Acute Hospital Care on Departure From the Emergency Department. Ann Emerg Med. 2019 Sep;74(3):345-356. doi: 10.1016/j.annemergmed.2019.04.012. Epub 2019 Jun 20. PMID 31229391
- [Background] Riddell M, Ospina M, Holroyd-Leduc JM. Use of Femoral Nerve Blocks to Manage Hip Fracture Pain among Older Adults in the Emergency Department: A Systematic Review. CJEM. 2016 Jul;18(4):245-52. doi: 10.1017/cem.2015.94. Epub 2015 Sep 10. PMID 26354332
- [Background] Ritcey B, Pageau P, Woo MY, Perry JJ. Regional Nerve Blocks For Hip and Femoral Neck Fractures in the Emergency Department: A Systematic Review. CJEM. 2016 Jan;18(1):37-47. doi: 10.1017/cem.2015.75. Epub 2015 Sep 2. PMID 26330019
- [Background] Akimoto T, Kobayashi T, Maita H, Osawa H, Kato H. Initial assessment of femoral proximal fracture and acute hip arthritis using pocket-sized ultrasound: a prospective observational study in a primary care setting in Japan. BMC Musculoskelet Disord. 2020 May 11;21(1):291. doi: 10.1186/s12891-020-03326-x. PMID 32393287
- [Background] Deleanu B, Prejbeanu R, Tsiridis E, Vermesan D, Crisan D, Haragus H, Predescu V, Birsasteanu F. Occult fractures of the proximal femur: imaging diagnosis and management of 82 cases in a regional trauma center. World J Emerg Surg. 2015 Nov 18;10:55. doi: 10.1186/s13017-015-0049-y. eCollection 2015. PMID 26587053
- [Background] Medero Colon R, Chilstrom ML. Diagnosis of an Occult Hip Fracture by Point-of-Care Ultrasound. J Emerg Med. 2015 Dec;49(6):916-9. doi: 10.1016/j.jemermed.2015.06.077. Epub 2015 Sep 26. PMID 26403984
- [Background] Pourmand A, Shokoohi H, Maracheril R. Diagnostic accuracy of point-of-care ultrasound in detecting upper and lower extremity fractures: An evidence-based approach. Am J Emerg Med. 2018 Jan;36(1):134-136. doi: 10.1016/j.ajem.2017.06.052. Epub 2017 Jun 27. No abstract available. PMID 28669695
- [Background] Schmid GL, Lippmann S, Unverzagt S, Hofmann C, Deutsch T, Frese T. The Investigation of Suspected Fracture-a Comparison of Ultrasound With Conventional Imaging. Dtsch Arztebl Int. 2017 Nov 10;114(45):757-764. doi: 10.3238/arztebl.2017.0757. PMID 29202925
- [Background] Chartier LB, Bosco L, Lapointe-Shaw L, Chenkin J. Use of point-of-care ultrasound in long bone fractures: a systematic review and meta-analysis. CJEM. 2017 Mar;19(2):131-142. doi: 10.1017/cem.2016.397. Epub 2016 Dec 5. PMID 27916021
- [Background] Landelijke Traumaregistratie 2018 - 2022, Landelijk Netwerk Acute zorg. Publicated September 2023.